CLINICAL TRIAL: NCT05101746
Title: Nitric Oxide Administration During Pediatric Cardiopulmonary Bypass Effects on End Organ Damage to the Brain and Kidney
Brief Title: Nitric Oxide Effect on Brain and Kidney in Pediatric Patients Undergoing Cardiopulmonary Bypass
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Bichell, Chief, Pediatric Cardiac Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211416
Record Dates: First submitted 2021-09-17; First posted 2021-11-01 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Congenital Heart Disease; Congenital Heart Defect; Congenital Heart Malformations
Keywords: pediatric heart surgery; congenital heart surgery
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitric oxide group (Experimental): Participants in this group will receive Nitric Oxide (NO) while undergoing Cardiopulmonary bypass (CPB)
  Interventions: Drug: Nitric Oxide (NO) 20 part per million (ppm)
- Standard of care cardiopulmonary bypass procedure (Active Comparator): Participants in this group will receive standard of care
  Interventions: Other: Standard of care cardiopulmonary bypass

INTERVENTIONS:
Drug: Nitric Oxide (NO) 20 part per million (ppm) — Nitric oxide will be mixed into the gas flow of the cardiopulmonary bypass (CPB) oxygenator, which will be kept at 1-3 L/min to allow for the desired NO delivery rate. NO levels will be maintained at 20ppm using a NO delivery system (INOmax, Mallinckrodt).
  Arms: Nitric oxide group
Other: Standard of care cardiopulmonary bypass — Cardiopulmonary bypass (CPB) will be performed using the departmental guidelines and standards. CPB will be performed using in a nonpulsatile flow with the System 1 Heart Lung Machine (Terumo Cardiovascular Systems, Ann Arbor, Mich). The maximum perfusion flow will be 200 ml/kg/minute. Blood pressure management will be selected based on the patient age and procedure. Temperature management will be to cool the patient 32 celsius (C).
  Arms: Standard of care cardiopulmonary bypass procedure

SUMMARY:
The goals of this study are:

1. To evaluate the neuroprotective effect of nitric oxide by measuring glial fibrillary acid protein (GFAP) before and after surgery. GFAP will be analyzed via an enzyme-linked immunosorbent assay (ELISA) kit. Patients will also be monitored post-operatively for delirium in the intensive care unit (ICU).
2. To evaluate the renal protective effect of nitric oxide by measuring neutrophil gelatinase-associated lipocalin (NGAL) before and after surgery. NGAL will also be analyzed via an ELISA kit. Patient creatinine will be monitored post-operatively.
3. To evaluate effect of nitric oxide on other ICU outcomes (invasive mechanical ventilation, days to extubation, ICU and hospital length of stay, and blood product administration).

DETAILED DESCRIPTION:
Corrective cardiac surgery for congenital heart disease (CHD) requiring cardiopulmonary bypass (CPB) is associated with numerous postoperative complications including neural tissue damage resulting in long-term neurocognitive deficits as well as acute kidney injury impacting renal function. Non-cardiac organ complications result in an increased mortality and length of hospital stay. Nitric oxide (NO) has been shown to play a protective role in a systemic inflammatory response, with administration of NO reducing damage to the liver, lungs, kidney, and brain in experimental models. Recent studies have demonstrated that for pediatric CHD patients undergoing corrective surgery administration of NO to the bypass circuit resulted in myocardial protection, reduced incidence of low cardiac output syndrome, and improved post-operative ICU course. NO in adult populations undergoing CPB has also been demonstrated to decrease the incidence of acute kidney injury.

Though prior studies have shown wide ranging protective effects from NO during CPB, these have not been fully characterized for neural and renal tissue for the pediatric population. Due to NO's promise in protective effects for other end organ damage the investigators are interested in investigating its potential to mitigate damage to neural and renal tissue. The investigators hypothesize that NO administration during CPB will be associated with reduced acute neurologic insult, reduced acute kidney injury postoperatively, and increased ventilator-free days.

To test these hypotheses the investigators propose a study where one group receives the current standard of care at Vanderbilt (standard surgery and CPB) and the other group receives NO administration during CPB in addition to standard surgery and CPB. The investigators propose using validated biomarkers to determine the effect of NO on the brain and kidney. GFAP is a biomarker for acute neurologic injury and NGAL is a biomarker of acute kidney injury. The biomarkers will be analyzed from blood drawn prior to and during surgery from existing lines in place as part of the procedure and will not necessitate additional needle sticks. No devices will be evaluated in this study; the investigators will only be measuring the effect of NO on neurological, renal and other ICU outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates and infants with CHD undergoing CPB for corrective surgery
2. Age <1 year old

Exclusion Criteria:

1. Requirement of inhaled NO immediately prior to surgery
2. Emergency surgery
3. Severe developmental delay at baseline defined as a score of ≥ 4 (severe disability) on the Pediatric Cerebral Performance Category (PCPC) Scale, referencing cognitive status prior to critical illness
4. Pre-existing renal disease
5. Inability to understand English or deafness that will preclude delirium evaluation. The inability to understand English in verbal participants will not result in exclusion when the research staff is proficient and/or translation services are actively available in that particular language.

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Level of glial fibrillary acid protein (GFAP) | baseline to peak rewarming temperature of blood (approximately 3 hours)
  GFAP will be measured via blood sample
Level of neutrophil gelatinase-associated lipocalin (NGAL) | baseline to 2 hours after CPB initiation (approximately 2 hours)
  NGAL will be measured via blood sample

SECONDARY OUTCOMES:
Daily prevalence of delirium as measured by preschool confusion assessment method for the ICU (psCAM-ICU) | date of admission to date of discharge from ICU (approximately 14 days)
  Daily prevalence of delirium will be monitored using the psCAM-ICU which is currently monitored daily in the pediatric ICU. The psCAM-ICU is designed to assess for delirium in critically ill children, with or without mechanical ventilation. The psCAM-ICU was designed with cognitive testing that is developmentally appropriate for infants-5 year olds.
  Patients are first assessed for arousal from -5 to +4 with -5 being unarousable to physical stimuli and +4 being combative. If arousal is greater than or equal to -3 than the patient is evaluated for the presence 4 features: 1) Acute change or fluctuating course of mental status, 2) Inattention, 3) Altered level of consciousness, 4) Disorganized thinking. Presence of 1 AND 2 AND either 3 OR 4 constitutes a positive result. The test results in the patient either being positive or negative for the presence of delirium.
Length of ICU stay | date of admission to date of discharge from ICU (approximately 14 days)
  intensive care unit (ICU) length of stay measured in days
Duration of mechanical ventilation | postoperative day 0 to hospital discharge (approximately 30 days)
  time spent on ventilator measured in days
Length of hospital stay | date of admission to date of hospital discharge (approximately 30 days)
  hospital length of stay measured in days
Mortality | date of admission to date of hospital discharge and/or 90 days post operation (approximately 90 days)
  In-hospital, 90-day mortality will be tracked and recorded
Organ dysfunction as measured by the pediatric Sequential Organ Failure Assessment | date of admission up to 14 days
  Organ dysfunctions will be tracked for up to 14 days during the Intervention Phase using the daily pediatric Sequential Organ Failure Assessment (pSOFA) scoring tool that is based on continuous as well as established predefined age appropriate cut offs for each organ failure. The following measurements are included: a. Creatinine (kidney), b. arterial oxygen saturation or arterial oxygen partial pressure over the fraction of inspired oxygen (lung), c. Total bilirubin (hepatic), d. Platelet count (coagulation), e. Glasgow coma score (neurologic), and f. Hemodynamic indices with +/-need for vasopressor (cardiovascular). These each receive a score of 0 to 4 based on the severity of the lab findings abnormality, with 0 being normal and 4 being the most severe. These are used to calculate a total score of 0 to 24, with 24 indicating a high risk of poor outcomes.
Functional Status | date of admission to date of hospital discharge (approximately 30 days)
  Functional Status Scale (FSS) will be measured at admission for baseline and again at hospital discharge. The FSS is a survey that tracks 6 domains (mental status, sensory, communication, motor function, feeding, respiratory) with a scoring from 1 to 5 each, with 1 being normal function and 5 being very severe dysfunction. Total scores will range from 6 to 30, with 6 being normal function and 30 being very severe dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: David P Bichell, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No